CLINICAL TRIAL: NCT04352998
Title: Effects of One Versus Two Doses of a Multi-Ingredient Pre-Workout Supplement on Metabolic Factors and Perceived Exertion During Moderate-Intensity Running in Females
Brief Title: Effects of a Multi-Ingredient Pre-Workout Supplement on Energy Expenditure During Running
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Illinois University (Other)
Collaborators: University of Wisconsin, La Crosse (Other); Mayo Clinic (Other); Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Clayton Camic, Associate Professor, Northern Illinois University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: NorthernIU
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Healthy
Keywords: caffeine; substrate utilization; thermogenic; fat oxidation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- One dose pre-workout supplement condition (Active Comparator): One dose/serving of a multi-ingredient pre-workout supplement was administered to the subjects.
  Interventions: Dietary Supplement: One dose pre-workout condition
- Two dose pre-workout supplement condition (Active Comparator): Two doses/servings of a multi-ingredient pre-workout supplement was administered to the subjects.
  Interventions: Dietary Supplement: Two dose pre-workout condition
- Placebo condition (Placebo Comparator): One dose/serving of a placebo was administered to the subjects.
  Interventions: Dietary Supplement: Placebo condition

INTERVENTIONS:
Dietary Supplement: One dose pre-workout condition — one dose of a multi-ingredient pre-workout supplement
  Arms: One dose pre-workout supplement condition
Dietary Supplement: Two dose pre-workout condition — two doses of a multi-ingredient pre-workout supplement
  Arms: Two dose pre-workout supplement condition
Dietary Supplement: Placebo condition — one dose of a placebo
  Arms: Placebo condition

SUMMARY:
The primary purpose of this study was to examine the acute effects of one versus two doses of a multi-ingredient pre-workout supplement on energy expenditure during moderate-intensity treadmill running. In addition, our second aim was to investigate the responses of associated metabolic factors (i.e. substrate utilization, measures of gas exchange), perceived exertion, and resting cardiovascular variables with one and two doses of the pre-workout supplement.

DETAILED DESCRIPTION:
This study utilized a randomized, double-blind, placebo-controlled, within-subjects crossover design (Figure 1). Each subject was required to visit the laboratory on five occasions with 72-96 hours between sessions. During the first laboratory visit, each subject performed an incremental test on a treadmill to familiarize the subjects with the testing procedures. For the second laboratory visit, each subject performed an incremental treadmill test to exhaustion to determine their ventilatory threshold (VT). The third laboratory visit was completed in the morning (06:00-09:00) and required subjects to consume a standardized meal after fasting overnight (8 hours) and sat quietly for 30 minutes before baseline heart rate and blood pressure values were recorded. The subjects were then randomly assigned to ingest the supplement (one or two doses) or placebo and sit quietly for another 30 minutes. The ingredients of the supplement (Cellucor, Bryan, TX) are provided in Table 1. The placebo was non-energetic and controlled for similar appearance and taste. At the 15-minute and 30-minute post-ingestion periods (of the pre-workout supplement or placebo), resting heart rate and blood pressure were recorded for a second and third time, respectively. Subjects then performed a 30-minute constant-velocity treadmill run at 90% of their VT. The subjects then returned to the laboratory for their fourth and fifth visits to ingest the remaining substances (1-dose, 2-dose, or placebo) and undergo the same testing procedures (including time of day) as the third visit. Each subject recorded 2-day food logs (MyFitnessPal, Inc., USA) prior to each laboratory visit.

ELIGIBILITY:
Inclusion Criteria:

* ran ≥ 16 km per week

Exclusion Criteria:

* (i) history of medical or surgical events, including cardiovascular disease, metabolic, renal, hepatic, or musculoskeletal disorders; (ii) use of any medication; (iii) use of nutritional supplements; (iv) habitual use of caffeine (≥ one cup of coffee or caffeinated beverage per day); or (v) participation in another clinical trial or investigation of another investigational product within 30 days prior to screening/enrollment.

Ages: 19 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2016-05-16 (Actual); Primary Completion 2016-05-16 (Actual); Study Completion 2016-05-16 (Actual)

PRIMARY OUTCOMES:
Energy expenditure | 30 minutes of exercise
  energy expenditure measured as kcals per minute

SECONDARY OUTCOMES:
substrate utilization | 30 minutes of exercise
  fat and carbohydrate oxidation
measures of gas exchange | 30 minutes of exercise
  oxygen consumption, respiratory exchange ratio
perceived exertion | 30 minutes of exercise
  ratings of perceived exertion (RPE)
resting cardiovascular variables | baseline and 30 minutes post-ingestion
  heart rate, systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Clayton Camic, PHD, Principal Investigator — Northern Illinois University

IPD SHARING:
Plan to Share IPD: No